CLINICAL TRIAL: NCT05329766
Title: A Phase 2 Trial to Evaluate the Safety and Efficacy of Combination Therapies in Patients With Advanced Upper Gastrointestinal Tract Malignancies (EDGE-Gastric)
Brief Title: A Safety and Efficacy Study of Treatment Combinations With and Without Chemotherapy in Adult Participants With Advanced Upper Gastrointestinal Tract Malignancies
Acronym: EDGE-Gastric
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARC-21; 2021-006291-16 (EudraCT Number); 2024-511917-40-00 (EU CTIS Number)
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-03

CONDITIONS: Gastrointestinal Tract Malignancies
Keywords: Domvanalimab; Quemliclustat; Zimberelimab; Esophageal adenocarcinoma; Gastric adenocarcinoma; Gastric cancer; Gastroesophageal junction cancer; Anti-PD-1 antibody; Anti-CD73; anti-TIGIT antibody
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Stomach Neoplasms | interventions — quemliclustat; zimberelimab; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- A1: First Line - Treatment Naïve Participants (Experimental): Domvanalimab and zimberelimab once every 4 weeks (Q4W) in addition to FOLFOX chemotherapy by intravenous (IV) infusion once every 2 weeks (Q2W)
  Interventions: Drug: Domvanalimab; Drug: Zimberelimab; Drug: Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin
- A2: First Line - Treatment Naïve Participants (Experimental): Zimberelimab Q4W in addition to chemotherapy with FOLFOX administered by IV infusion Q2W
  Interventions: Drug: Zimberelimab; Drug: Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin
- A3 First Line - Treatment Naïve Participants (Experimental): Non-randomized A3 safety run-in cohort: Domvanalimab and zimberelimab co-administered Q4W via IV infusion over 60 minutes in addition to FOLFOX chemotherapy via IV infusion Q2W.
  After completion of A3 safety run-in cohort, participants are randomized to the A3 arm. Domvanalimab and zimberelimab co-administered Q4W via IV infusion over 30 minutes, in addition to FOLFOX chemotherapy via IV infusion Q2W
  Interventions: Drug: Domvanalimab; Drug: Zimberelimab; Drug: Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin
- A4 First Line - Treatment Naïve Participants (Experimental): Zimberelimab administered Q4W via IV infusion over 30 minutes, in addition to FOLFOX chemotherapy via IV infusion Q2W
  Interventions: Drug: Zimberelimab; Drug: Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin
- B1: Second Line or greater Checkpoint Inhibitor Naïve Participants (Experimental): Domvanalimab and zimberelimab administered once every three weeks (Q3W) by IV infusion
  Interventions: Drug: Domvanalimab; Drug: Zimberelimab
- B2: Second Line or greater Checkpoint Inhibitor Naïve Participants (Experimental): Quemliclustat Q2W and zimberelimab Q4W administered by IV infusion
  Interventions: Drug: Quemliclustat; Drug: Zimberelimab
- Cohort C1: Second Line or greater - Checkpoint Inhibitor Experienced Participants (Experimental): Domvanalimab and zimberelimab Q3W administered by IV infusion
  Interventions: Drug: Domvanalimab; Drug: Zimberelimab

INTERVENTIONS:
Drug: Domvanalimab — Administered as specified in the treatment arm
  Arms: A1: First Line - Treatment Naïve Participants; A3 First Line - Treatment Naïve Participants; B1: Second Line or greater Checkpoint Inhibitor Naïve Participants; Cohort C1: Second Line or greater - Checkpoint Inhibitor Experienced Participants
Drug: Quemliclustat — Administered as specified in the treatment arm
  Arms: B2: Second Line or greater Checkpoint Inhibitor Naïve Participants
Drug: Zimberelimab — Administered as specified in the treatment arm
Drug: Fluorouracil — Administered as specified in the treatment arm
  Arms: A1: First Line - Treatment Naïve Participants; A2: First Line - Treatment Naïve Participants; A3 First Line - Treatment Naïve Participants; A4 First Line - Treatment Naïve Participants
Drug: Leucovorin — Administered as specified in the treatment arm
  Arms: A1: First Line - Treatment Naïve Participants; A2: First Line - Treatment Naïve Participants; A3 First Line - Treatment Naïve Participants; A4 First Line - Treatment Naïve Participants
Drug: Oxaliplatin — Administered as specified in the treatment arm
  Arms: A1: First Line - Treatment Naïve Participants; A2: First Line - Treatment Naïve Participants; A3 First Line - Treatment Naïve Participants; A4 First Line - Treatment Naïve Participants

SUMMARY:
The purpose of this study is to evaluate the safety and preliminary clinical activity of treatment combinations with and without chemotherapy in participants with locally advanced unresectable or metastatic gastric, GEJ, and esophageal adenocarcinoma. Chemotherapy will consist of FOLFOX (oxaliplatin, leucovorin, fluorouracil).

ELIGIBILITY:
Key Inclusion Criteria:

* Participants with histologically confirmed diagnosis of locally advanced unresectable or metastatic gastric, GEJ, or esophageal adenocarcinoma with life expectancy ≥3 months as assessed by the Investigator
* Eastern cooperative oncology group (ECOG) Performance Score of 0-1
* At least one measurable target lesion per RECIST v1.1.
* Adequate organ and marrow function
* Able to provide an archival tumor sample that is representative of the cancer under investigation and suitable for central PD-L1 testing

Key Exclusion Criteria:

* Participants with underlying medical conditions that, in the Investigator's or Sponsor's opinion, will make the administration of investigational products hazardous
* Only for Cohort A: Known Human Epidermal Growth Factor Receptor 2 (HER-2) positive tumor
* Known untreated, symptomatic, or actively progressing central nervous system (brain) metastases. Participants with leptomeningeal metastases are excluded from enrollment.
* Discontinued use of prior immune checkpoint therapy due to immune related adverse events; received prior treatment with an anti-TIGIT monoclonal antibody.
* History of trauma or major surgery within 28 days prior to enrollment.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to 18 months
Objective Response Rate (ORR) as measured by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to 18 months

SECONDARY OUTCOMES:
Objective Response Rate (ORR) as measured by PD-L1 Expression Level | Up to 18 months
Overall survival (OS) | From date of first dose until the date of death due to any cause (approximately 18 months)
Progression-free survival (PFS) as determined by the Investigator according to RECIST v1.1 | Up to 18 months
Disease Control (complete response, partial response, or stable disease) for greater than equal to 12 weeks | Up to 18 months
Duration of response (DOR) as determined by the Investigator according to RECIST v1.1 | Up to 18 months
Plasma concentration of domvanalimab | Up to 18 months
Plasma concentration of zimberelimab | Up to 18 months
Plasma concentration of quemliclustat | Up to 18 months
Percentage of participants with anti-drug antibodies to domvanalimab | Up to 18 months
Percentage of participants with anti-drug antibodies to zimberelimab | Up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Arcus Biosciences, Inc.
Locations (49):
- United States (16):
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Santa Monica, California
  - Yale Cancer Center, Derby, Connecticut
  - Florida Cancer Specialist - South, Fort Myers, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Florida Cancer Specialist - North, St. Petersburg, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Columbia University, New York, New York
  - Duke University, Durham, North Carolina
  - Zangmeister Cancer Center, Columbus, Ohio
  - OU - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - SCRI Tennessee Oncology - Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Virginia Cancer Specialists, Fairfax, Virginia
- UHN - Princess Margaret Cancer Centre, Toronto, Canada
- Chile (4):
  - Clínica San Carlos de Apoquindo, Las Condes
  - Bradford Hill Centro de Investigaciones Clinicas, Recoleta
  - Centro de Estudios Clínicos SAGA, Santiago
  - Clínica Universidad Católica del Maule, Talca
- France (11):
  - Institut Bergonié _ Bordeaux, Bordeaux
  - CHU de Brest_Brest, Brest
  - Centre Baclesse - CAEN, Caen
  - Centre Oscar Lambret _ LILLE, Lille
  - Centre Léon Bérard _ Lyon, Lyon
  - Hôpital Timone - Marseille, Marseille
  - Institut de Recherche en Cancerologie de Montpellier, Montpellier
  - Centre Armoricain de Radiothérapie, d'Imagerie Médicale et d'Oncologie, Plérin
  - Pôle Régional de Cancérologie - Service d'Oncologie Médicale - Poitiers, Poitiers
  - CHU de Toulouse_Oncopole, Toulouse
  - Gustave Roussy - Villejuif, Villejuif
- Serbia (5):
  - MSB - Medicinski Sistem Beograd, Belgrade
  - University Clinical Center of Serbia, Belgrade
  - University Hospital Medical Center (KBC) Bezanijska Kosa, Belgrade
  - Institute of Oncology of Vojvodina, Kamenitz
  - Clinical Center Kragujevac, Kragujevac
- South Korea (12):
  - Dong-A University Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Chonnam National University Hwasun Hospital, Hwasun
  - CHA Bundang Medical Center, Seongnam-si
  - Asan Medical Center Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital Cancer Center, Seoul
  - Ajou University Hospital, Suwon
  - St. Vincent's Hospital, The Catholic University of Korea, Suwon

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents (e.g., protocol, Statistical Analysis Plan [SAP], Clinical Study Report [CSR]) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
  For more information, please visit our website.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy

REFERENCES:
- [Derived] Janjigian YY, Oh DY, Pelster M, Wainberg ZA, Prusty S, Nelson S, DuPage A, Thompson A, Koralek DO, Sison EAR, Rha SY. Domvanalimab and zimberelimab in advanced gastric, gastroesophageal junction or esophageal cancer: a phase 2 trial. Nat Med. 2025 Dec;31(12):4274-4280. doi: 10.1038/s41591-025-04022-w. Epub 2025 Oct 18. PMID 41109921
- See also: ARC-21 - Public website — https://trials.arcusbio.com/study/?id=ARC-21